CLINICAL TRIAL: NCT03889327
Title: Intervention to Reduce Distress from Perceived Cognitive Impairment in Multiple Sclerosis
Brief Title: Intervention to Reduce Perceived Cognitive Impairment in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: University of Kansas (Other)
Responsible Party: Principal Investigator, Jared Bruce, Professor, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-180
Record Dates: First submitted 2018-03-12; First posted 2019-03-26 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2020-11

CONDITIONS: Multiple Sclerosis
Keywords: Perceived Cognitive Impairment; Neuropsychology
MeSH Terms: conditions — Multiple Sclerosis | interventions — Health

STUDY DESIGN:
Intervention Model Description: Once written consent is obtained, patients will complete baseline self-report questionnaires and neuropsychological tests. Immediately following the baseline assessment, patients will be notified of their eligibility. If inclusion criteria is met, patients will be randomized, based on gender in a 2, 4, or 6 block randomization into either the treatment or control group. Patients and the research investigator will be blind to treatment assignment. Participants will complete the intervention and follow-up questionnaires through the research electronic data capture (REDCap), a secure internet-based computerized system. The REDCap link will be emailed to participants within 24 hours of their enrollment into the study. Participants should initiate the intervention at their earliest convenience. The one-week post-intervention follow-up questionnaires will also be emailed directly to participants, and accessed using a REDCap link.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 2, 4, and 6 blocked randomization (by gender) was conducted via computer generator. Group assignment was specified and sealed in individual envelopes by a study coordinator who is not involved in the current project. After participants are enrolled and complete the baseline evaluation, the appropriate envelope will be selected, based on gender, containing group assignment, and the subsequent intervention will be administered. Group assignment is not established until after the baseline evaluation has been conducted. Determining randomization will take place at a separate location from the recruitment/baseline site. No study member will have direct contact with participants following the baseline evaluation since the intervention is computerized and replies on emailing the study link to complete the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Feedback and Psychoeducation (CFP) (Experimental): Participants assigned to the cognitive feedback and psychoeducation (CFP) treatment group will watch a brief video integrating both neuropsychological test feedback and psychoeducation. The computerized intervention will cover MS disease-related information, define objective cognition, explain neuropsychological assessment, and inform patients of their cognitive test performance outcomes. The CFP intervention will also define and explain perceived cognition and subjective measures of cognition, and compare objective performance on neuropsychological tests to a subjective measure of perceived cognition. The intervention will also discuss emotion, attention, and misattribution related to PCI. The proposed intervention will incorporate expert testimony on MS disease course and related symptomology and interpretations of neuropsychological test performance.
  Interventions: Behavioral: Neuropsychological Feedback & Psychoeducation (Cognition)
- Healthy Eating Habits (HEH) (Active Comparator): The control group, healthy eating habits (HEH) group, will watch a brief psychoeducational video of same length in time as the treatment group. The control intervention will include information on importance of healthy eating habits and benefits of a healthy diet including medical outcomes such as reduced blood pressure, and decreased risk of stroke and cardiovascular disease. This intervention will also cover recommended serving sizes for daily helpings of fruits and vegetables, and ways to incorporate fruits and vegetables into meals throughout the day. The proposed control intervention will include expert testimony from a nutritionist and expert dietician.
  Interventions: Behavioral: Psychoeducation (Health)

INTERVENTIONS:
Behavioral: Neuropsychological Feedback & Psychoeducation (Cognition) — The customary practice of providing feedback on neuropsychological test performance can address patient misperceptions of cognitive impairment by distinguishing between perceived and objective neuropsychological test performance. Explaining how normative data is derived by comparison to same age peers, patients are able to better understand their current cognitive functioning. The proposed intervention will employ both psychoeducation and neuropsychological feedback for participants assigned to the treatment group, and psychoeducation for participants assigned to the control group. Both groups will watch 3 brief videos (exactly the same length in time) and answer two qualitative questions following each video.
  Arms: Cognitive Feedback and Psychoeducation (CFP)
Behavioral: Psychoeducation (Health) — Information on importance of healthy eating habits and benefits of a healthy diet including medical outcomes such as reduced blood pressure, and decreased risk of stroke and cardiovascular disease. This intervention will also cover recommended serving sizes for daily helpings of fruits and vegetables, and ways to incorporate fruits and vegetables into meals throughout the day. The control intervention will include expert testimony from a nutritionist and expert dietician.
  Arms: Healthy Eating Habits (HEH)

SUMMARY:
Multiple sclerosis (MS) is among the most prevalent autoimmune diseases among young and middle-aged adults. Up to 65% of MS patients experience objective cognitive impairment including problems with information processing speed, memory, and executive functioning. However, patients commonly overestimate the extent of their cognitive dysfunction which can result in inaccurate perceptions of their true cognitive abilities. Exaggerated perceptions of cognitive impairment are predictive of future decline and associated with depression, anxiety, and reduced quality of life. Despite this, no study has examined an intervention aimed at changing misperceptions related to perceived cognitive impairment in MS when objective measures are incongruent with self-reported cognitive symptoms. The purpose of the present study is to develop and pilot a brief intervention for MS patients who perceive cognitive impairment, but perform in the normal or expected range on objective measures of cognition.

DETAILED DESCRIPTION:
Concern over worsening cognitive functioning has been shown to significantly impact patients' lives. More than half of all MS patients demonstrate clinically significant cognitive dysfunction, making it one of the leading causes of disability in MS. Cognitive deficits often manifest in areas associated with information processing speed, memory, and executive functioning. Resulting sequela can have profound implications on employment, interpersonal relationships, and activities of daily living. Despite the prevalence of cognitive dysfunction in MS, most studies find little to no relationship between perceived and objective cognition in MS. Research shows that some patients overestimate the extent of their cognitive deficits. PCI is associated with poor self-efficacy, social, and occupational difficulties. Evidence suggests that negative emotional states may contribute to overestimated PCI in MS. Exaggerated perceptions of impaired cognition may be intensified by the presence of other MS symptoms, which can affect the way patients report disease activity to healthcare providers and complicate detection of relevant disease symptomatology.

Overestimating cognitive impairment has been observed in other patient populations, but it is especially problematic in MS and can provide an opportunity to inform patients about discrepancies between perceived and objective cognitive functioning. Since physicians spend significant amounts of time negating unsubstantiated healthcare concerns, an intervention aimed at decreasing PCI in MS may improve long-term healthcare outcomes as well as the quality of time that physicians spend with patients. Neuropsychological test results can be used as objective evidence against perceived cognitive impairment to change patients perceptions, if conveyed in an appropriate and nonthreatening manner.

Educating patients about the influence of emotional dysfunction and misattribution as it relates to PCI may also decrease concern regarding cognitive decline and MS. Specifically, internal processes such as emotional dysfunction, including a globally negative world view can increase dissociative experiences that cause patients to misattribute normal cognitive errors as MS-related cognitive decline. This model may inform patients understanding of medically unsubstantiated PCI, allowing them to consider alternative factors associated with common cognitive errors aside from MS.

Although many studies have aimed to improve cognition in MS through pharmacological treatments, cognitive rehabilitation, and psychotherapy, to the investigators knowledge, this is the first study to examine a psychoeducational intervention to decrease exaggerated perceptions of cognitive impairment in MS. For the present study, the investigators will develop a brief computer-based intervention for MS patients who perceive cognitive decline incongruent with objective measures of cognition. The proposed intervention will incorporate feedback from neuropsychological tests, including comparisons of perceived and objective performance. The intervention will also introduce psychoeducation about causes of PCI, such as emotional distress, attention, and misattribution. It is hoped that by combining neuropsychological test feedback and psychoeducation, patients may better understand differences between perceived and objective cognition, which in turn, may reduce concern and offer alternative explanations for PCI.

Goals and Hypotheses

For the current study, the investigators will develop a brief computer-based intervention for MS patients who perceive cognitive decline that is incongruent with objective measures of cognitive functioning. The project will accomplish the following specific aims:

1. Develop and assess the feasibility and acceptability of a brief, single-session, computerized intervention (cognitive feedback and psychoeducation; CFP) as part of a randomized controlled pilot trial to reduce perceived cognitive impairment and distress associated with perceived cognitive impairment that is incongruent with objective measures of cognition in MS patients.
2. Examine whether the intervention reduces distress related to perceived cognitive deficits. The investigators hypothesize that patients in the CFP group will report less distress over perceived cognitive impairment compared to the control group immediately after and one week following the intervention.
3. Examine patients understanding of factors that contribute to perceived and objective cognitive impairment in MS. The investigators hypothesize that patients in the CFP group will have an increased understanding of the role that negative emotion, misattribution, and other secondary factors play in the formation of perceived cognitive deficits when compared to patients assigned to the HEH group.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MS by a board-certified neurologist
* a total score > 40 on the Perceived Deficits Questionnaire (PDQ) based on previous research that identifies this cutoff score as clinically significant in the MS population and two standard deviations below average in the general population (Ruth Ann Marrie, Gordon J. Chelune, Deborah M. Miller, & Jeffrey A. Cohen, 2005)
* score in the low average or better range on the Wechsler Test of Adult Reading (WTAR)
* average score equal to or greater than the 16th percentile on the Hopkins Verbal Learning Test (HVLT), Symbol Digit Modalities Test (SDMT), Controlled Oral Word Association Test (COWAT), and Wisconsin Card Sorting Task (WCST)
* average T score on the HVLT, SDMT, COWAT, and WCST no more than one standard deviation below the WTAR T score
* access to a computer and a personal email account
* English-speaking

Exclusion Criteria:

* no severe sensory, motor, physical, or neurological impairment that would make participation in the study insurmountable
* no history of nervous system disorder other than MS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Feasibility and Acceptability Questionnaire | 5 minutes
  All participants complete a feasibility and acceptability questionnaire upon study completion. The questionnaire will address satisfaction with study participation, effectiveness and convenience of the intervention, and short answer questions on newly acquired information, application of information learned, and feelings about the new information. Participants will also be asked if they perceived the intervention as helpful and if they would be willing to recommend it to other MS patients. This measure will be scored quantitatively, ranging from 0-85 possible points, where higher scores indicated greater feasibility and acceptability of the intervention.

SECONDARY OUTCOMES:
Cognition Quiz | 5 minutes
  Examine patients understanding of factors that contribute to perceived and objective cognitive impairment in MS. All participants will complete the cognition quiz. Scores range from 0-21, where higher scores indicated greater knowledge of perceived and objective cognition. Within participant analysis will be used to compare changes in score from baseline to immediate post intervention.
Perceived Cognitive Impairment-Distress (PCI-D) | 5 minutes
  Examine distress related to perceived cognitive deficits. Within subject comparisons will be made, examining baseline and immediate post intervention responses on this questionnaire. Scores range from 0-60, higher scores indicate greater distress over perceived cognitive deficits.

CONTACTS AND LOCATIONS:
Overall Officials: Jared Bruce, PhD, Study Chair — UMKC Faculty
Locations (1):
- University of Kansas Department of Neurology, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amato MP, Ponziani G, Rossi F, Liedl CL, Stefanile C, Rossi L. Quality of life in multiple sclerosis: the impact of depression, fatigue and disability. Mult Scler. 2001 Oct;7(5):340-4. doi: 10.1177/135245850100700511. PMID 11724451
- [Background] Kujala P, Portin R, Ruutiainen J. The progress of cognitive decline in multiple sclerosis. A controlled 3-year follow-up. Brain. 1997 Feb;120 ( Pt 2):289-97. doi: 10.1093/brain/120.2.289. PMID 9117376
- [Background] Beier M, Amtmann D, Ehde DM. Beyond depression: Predictors of self-reported cognitive function in adults living with MS. Rehabil Psychol. 2015 Aug;60(3):254-62. doi: 10.1037/rep0000045. Epub 2015 Jul 20. PMID 26192051
- [Background] Benedict RH, Cookfair D, Gavett R, Gunther M, Munschauer F, Garg N, Weinstock-Guttman B. Validity of the minimal assessment of cognitive function in multiple sclerosis (MACFIMS). J Int Neuropsychol Soc. 2006 Jul;12(4):549-58. doi: 10.1017/s1355617706060723. PMID 16981607
- [Background] Olazaran J, Cruz I, Benito-Leon J, Morales JM, Duque P, Rivera-Navarro J. Cognitive dysfunction in multiple sclerosis: methods and prevalence from the GEDMA Study. Eur Neurol. 2009;61(2):87-93. doi: 10.1159/000177940. Epub 2008 Nov 28. PMID 19039226
- [Background] Kinsinger SW, Lattie E, Mohr DC. Relationship between depression, fatigue, subjective cognitive impairment, and objective neuropsychological functioning in patients with multiple sclerosis. Neuropsychology. 2010 Sep;24(5):573-80. doi: 10.1037/a0019222. PMID 20804245
- [Background] Benedict RH. Effects of using same- versus alternate-form memory tests during short-interval repeated assessments in multiple sclerosis. J Int Neuropsychol Soc. 2005 Oct;11(6):727-36. doi: 10.1017/S1355617705050782. PMID 16248908
- [Background] Bruce JM, Bruce AS, Hancock L, Lynch S. Self-reported memory problems in multiple sclerosis: influence of psychiatric status and normative dissociative experiences. Arch Clin Neuropsychol. 2010 Feb;25(1):39-48. doi: 10.1093/arclin/acp092. Epub 2009 Dec 3. PMID 19959565
- [Background] Kalmar JH, Gaudino EA, Moore NB, Halper J, Deluca J. The relationship between cognitive deficits and everyday functional activities in multiple sclerosis. Neuropsychology. 2008 Jul;22(4):442-9. doi: 10.1037/0894-4105.22.4.442. PMID 18590356
- [Background] Rao SM, Leo GJ, Ellington L, Nauertz T, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. II. Impact on employment and social functioning. Neurology. 1991 May;41(5):692-6. doi: 10.1212/wnl.41.5.692. PMID 1823781
- [Background] Basso MR, Shields IS, Lowery N, Ghormley C, Combs D, Arnett PA, Johnson J. Self-reported executive dysfunction, neuropsychological impairment, and functional outcomes in multiple sclerosis. J Clin Exp Neuropsychol. 2008 Nov;30(8):920-30. doi: 10.1080/13803390801888733. PMID 18608679
- [Background] Middleton LS, Denney DR, Lynch SG, Parmenter B. The relationship between perceived and objective cognitive functioning in multiple sclerosis. Arch Clin Neuropsychol. 2006 Aug;21(5):487-94. doi: 10.1016/j.acn.2006.06.008. Epub 2006 Aug 1. PMID 16879944
- [Background] Akbar N, Honarmand K, Feinstein A. Self-assessment of cognition in Multiple Sclerosis: the role of personality and anxiety. Cogn Behav Neurol. 2011 Sep;24(3):115-21. doi: 10.1097/WNN.0b013e31822a20ae. PMID 21904202
- [Background] Akbar N, Honarmand K, Kou N, Feinstein A. Validity of a computerized version of the symbol digit modalities test in multiple sclerosis. J Neurol. 2011 Mar;258(3):373-9. doi: 10.1007/s00415-010-5760-8. Epub 2010 Oct 6. PMID 20924594
- [Background] Cull A, Hay C, Love SB, Mackie M, Smets E, Stewart M. What do cancer patients mean when they complain of concentration and memory problems? Br J Cancer. 1996 Nov;74(10):1674-9. doi: 10.1038/bjc.1996.608. PMID 8932354
- [Background] Sawrie SM, Martin RC, Kuzniecky R, Faught E, Morawetz R, Jamil F, Viikinsalo M, Gilliam F. Subjective versus objective memory change after temporal lobe epilepsy surgery. Neurology. 1999 Oct 22;53(7):1511-7. doi: 10.1212/wnl.53.7.1511. PMID 10534260
- [Background] Sawrie SM, Marson DC, Boothe AL, Harrell LE. A method for assessing clinically relevant individual cognitive change in older adult populations. J Gerontol B Psychol Sci Soc Sci. 1999 Mar;54(2):P116-24. doi: 10.1093/geronb/54b.2.p116. PMID 10097774
- [Background] van Gorp WG, Satz P, Hinkin C, Selnes O, Miller EN, McArthur J, Cohen B, Paz D. Metacognition in HIV-1 seropositive asymptomatic individuals: self-ratings versus objective neuropsychological performance. Multicenter AIDS Cohort Study (MACS). J Clin Exp Neuropsychol. 1991 Sep;13(5):812-9. doi: 10.1080/01688639108401091. PMID 1955533
- [Background] Maor Y, Olmer L, Mozes B. The relation between objective and subjective impairment in cognitive function among multiple sclerosis patients--the role of depression. Mult Scler. 2001 Apr;7(2):131-5. doi: 10.1177/135245850100700209. PMID 11424633
- [Background] Arnett PA, Rao SM, Grafman J, Bernardin L, Luchetta T, Binder JR, Lobeck L. Executive functions in multiple sclerosis: an analysis of temporal ordering, semantic encoding, and planning abilities. Neuropsychology. 1997 Oct;11(4):535-44. doi: 10.1037//0894-4105.11.4.535. PMID 9345697
- [Background] Mittenberg W, Canyock EM, Condit D, Patton C. Treatment of post-concussion syndrome following mild head injury. J Clin Exp Neuropsychol. 2001 Dec;23(6):829-36. doi: 10.1076/jcen.23.6.829.1022. PMID 11910547
- [Background] Bruce JM, Bruce AS, Arnett PA. Response variability is associated with self-reported cognitive fatigue in multiple sclerosis. Neuropsychology. 2010 Jan;24(1):77-83. doi: 10.1037/a0015046. PMID 20063948
- [Background] Carone DA. But the Scores Don't Show How I Really Function: A Feedback Method to Reveal Cognitive Distortions Regarding Normal Neuropsychological Test Performance. Appl Neuropsychol Adult. 2017 Mar-Apr;24(2):160-168. doi: 10.1080/23279095.2015.1116074. Epub 2016 Apr 4. PMID 27045631